CLINICAL TRIAL: NCT07295314
Title: Effect of Antifungals on the Intestinal Microbiome - a Randomized, Controlled, Proof-of-concept Trial
Acronym: FAME
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, W. J. Wiersinga, MD, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.0143
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gut Microbiome; Healthy Adult Male; Antifungal Therapy
Keywords: Fluconazole; Antifungal Drugs; Mycobiome; Bacteriome; Microbiota Diversity; Innate Immune Response; Healthy Volunteers
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive fluconazole or no intervention in a parallel-group design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluconazole (Experimental): Participants will receive oral fluconazole 200mg once daily for 14 days.
  Interventions: Drug: Fluconazole 200mg tab
- No Intervention (No Intervention): Participants assigned to the control arm will not receive any treatment.

INTERVENTIONS:
Drug: Fluconazole 200mg tab — Oral administration of one 200 mg fluconazole tablet once daily for 14 days.
  Arms: Fluconazole

SUMMARY:
The goal of this clinical trial is to learn how the antifungal drug fluconazole affects the gut microbiome and immune system in healthy volunteers.

The main questions it aims to answer are:

* Does fluconazole change the gut bacteriome and mycobiome composition after 14 days of treatment?
* How long do these changes last (4 weeks and 6 months after treatment)?
* Does fluconazole affect the body's immune responses, such as blood cell activity and antifungal antibodies?

Researchers will compare two groups: participants who take fluconazole for 14 days and participants who receive no intervention.

Participants will:

* Either take one fluconazole tablet (200 mg) daily for 14 days, or receive no treatment
* Provide stool samples and blood samples at several timepoints
* Return for follow-up visits up to 6 months after treatment

This study is conducted at Amsterdam UMC, location AMC, with a planned enrollment of 50 healthy male volunteers aged 18-35 years.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-35 years of age at the time of signing informed consent
* Healthy, as determined by medical history and physical examination; minor clinical abnormalities allowed if not introducing additional risk or interfering with study procedures
* Capable of giving written informed consent and able to comply with study requirements
* Normal defecation pattern (≤3 times/day and ≥3 times/week)

Exclusion Criteria:

* Major illness in the past 3 months, or significant chronic medical illness deemed unfavorable for enrollment
* Past or current gastrointestinal disease that may influence the gut microbiota (including inflammatory bowel disease or medication-treated irritable bowel syndrome)
* History of immunodeficiency
* History of malignancy
* Alcohol intake >3 units/day on average
* Known allergy to antifungal drugs
* Use of antibiotics (except topical) within the past 3 months
* Use of antifungals (except topical) within the past 3 months
* Planned prolonged travel (>4 weeks) to tropical countries during the study period
* Receipt of an investigational product within 3 months prior to study day 0
* Use of prescription or non-prescription drugs, herbal or dietary supplements within 3 months (unless deemed safe by investigator)
* Difficulty with blood donation or poor venous access in either arm
* Donation of >500 mL of blood in the past 3 months
* Any other condition or circumstance that, in the investigator's opinion, could be harmful to the subject or compromise data interpretation

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy males are eligible to participate.
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Effect of fluconazole on the intestinal microbiome | 14 days (end of treatment)
  Difference in gut bacteriome and mycobiome composition, ⍺- and ß-diversity between adults treated with an antifungal (fluconazole) and no intervention directly after completion of antifungal treatment (t=14 days).

SECONDARY OUTCOMES:
Gut microbiome and mycobiome composition at 6 months post-treatment | 6 months post-treatment
  Differences in gut bacteriome and mycobiome composition, including α- and β diversity, between fluconazole and no-intervention arms and compared to baseline, 6 months after completion of fluconazole treatment.
Gut microbial functional profiles after fluconazole treatment | Baseline, 14 days, 4 weeks, and 6 months
  Differences in gut microbial functional profiles, including metabolic pathways and in vitro fecal microbial fermentation, between fluconazole and no-intervention arms
Systemic innate immune responses after fluconazole treatment | Baseline, 14 days, 4 weeks, and 6 months
  Differences in host systemic innate immune response profiles between fluconazole and no-intervention arms at baseline, 14 days, 4 weeks, and 6 months. Responses will be assessed using ex vivo stimulation assays of peripheral blood mononuclear cells and neutrophils, and measurement of antifungal antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No